CLINICAL TRIAL: NCT00181506
Title: HI-CHART: A Phase I/II Study on the Feasibility of High-Dose Accelerated Conformal Radiotherapy in Patients With Inoperable Non-Small Cell Lung Cancer.
Brief Title: HI-CHART:Feasibility of High-Dose Accelerated Conformal Radiotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01.1314L; MEC MAASTRO clinic: 0105
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: radiotherapy; radiation dose; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

INTERVENTIONS:
Procedure: dose escalation (radiotherapy treatment schedule)

SUMMARY:
In this study we try to increase the radiation dose, while reducing or keeping the radiation schedule below 4 weeks.

The study hypothesis is that it is feasible to administer hyperfractionated accelerated radiotherapy to patients with inoperable or locally advanced non small cell lung cancer.

DETAILED DESCRIPTION:
Non-small cell lung cancer is still the most common cancer and the main cause of cancer death. Treatment of choice for these patients is often radiotherapy, which results in an overall 5-year survival rate between 5 and 10%. The addition of chemotherapy improves survival by a few percentages and is therefore considered standard treatment for patients with stage III disease.

However, several factors have been identified that have an impact on the local control but also on survival.

1. There is a dose-effect relationship. A higher dose results in a better survival rate. However, higher radiation doses are currently not delivered with conventional radiation due to the tolerance of normal tissue.
2. The time factor plays an important role in radiotherapy. Prolonging the overall treatment time decreases the outcome of radiotherapy. Radiobiological modelling of data shows that the overall treatmetn time (OTT) should be kept below 4 weeks. Results from studies support this conclusion.

So, probably the best results will be achieved when a very high radiation dose can be delivered within 4 weeks, without severally damaging normal tissue.

In order to achieve this goal, an hyperfractionated accelerated treatment regimen together with a technically very advanced radiation technique to avoid as much normal tissue as possible, will be used in this study.

ELIGIBILITY:
Inclusion Criteria:

histological or cytological diagnosis of non-small cell lung cancer stage I-III disease, except supra-clavicular lymph nodes availability for participating in the detailed follow-up of the protocol able to tolerate a radiation course according to the protocol guidelines in case of previous chemotherapy, radiotherapy can start after a minimum of 3 weeks after the last CT course good performance status: Karnofsky>=70%, WHO performance status 0-2 adequate lung functions allowing the radiation according to the guidelines protocol no severe recent cardiac disease absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; conditions should be discussed with the patient before registration in the trial -

Exclusion Criteria:

patients who have a peripherally located lower lobe tumor and contralateral upper mediastinal nodes malignant pleural or pericardial effusion concurrent chemotherapy programs history of a prior malignancy excluding non melanoma skin cancer or in-situ cancer history of prior chest irradiation recent myocardial infraction uncontrolled infectious disease distant metastases (stage IV)

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2001-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
acute toxicity

SECONDARY OUTCOMES:
late toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Rinus Wanders, MD, Principal Investigator — Maastricht Radiation Oncology (MAASTRO clinic)
Locations (1):
- Maastircht Radiation Oncology, Heerlen, Limburg, Netherlands